CLINICAL TRIAL: NCT07092774
Title: Real-World Safety and Effectiveness of Catheter Ablation of Paroxysmal Atrial Fibrillation as Initial Rhythm Control Therapy With the THERMOCOOL SMARTTOUCH SF Catheter - A Sub-study of REAL AF Registry
Brief Title: Real-world Safety and Effectiveness Registry of Catheter Ablation of Paroxysmal Atrial Fibrillation as Initial Control Therapy With the Thermocool SmartTouch SF Catheter (A Sub-study of REAL AF Registry)
Acronym: First Line
Status: Active, not recruiting | Type: Observational
Sponsor: Heart Rhythm Clinical and Research Solutions, LLC (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BWI-CS-004-F
Record Dates: First submitted 2025-07-22; First posted 2025-07-30 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Paroxysmal Atrial Fibrillation (PAF)
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Ablation — Ablation procedure using the Thermocool Smarttouch SF

SUMMARY:
To generate real-world evidence from the parent study, REAL AF registry, on the use of Thermocool SmartTouch SF (STSF) catheter in ablation for the treatment of paroxysmal atrial fibrillation (PAF).

DETAILED DESCRIPTION:
The primary objective of this registry is to evaluate effectiveness and safety of Thermocool STSF catheter to support an indication extension of the STSF catheter using real world data from the REAL AF registry. Subjects included in the registry will be those in which the STSF catheter is used for the treatment of symptomatic PAF in antiarrhythmic drug (AAD) naive patients as an initial rhythm control therapy. The registry will involve retrospective analysis of data prospectively collected from the REAL AF registry. The registry will include consecutive, eligible patients from the REAL AF registry, starting from October 2021 who meet the sub-study eligibility criteria until 344 eligible subjects are identified. Eligible patients from all participating centers in the REAL AF registry will be included, except for sites with standard-of-care rhythm monitoring less than 48 hours and those that do not perform 6-12 month follow up as standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with symptomatic PAF
* First time ablation
* Ablation performed with the Thermocool STSF catheter
* Age 18 or over at the time of the index ablation procedure

Exclusion Criteria:

* Received Class I or III antiarrhythmic drug prior to the index ablation.
* Did not previously consent for their anonymized data to be used for research purposes.
* Rhythm monitoring less than 48 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sub-study population will consist of Class I/III AAD naïve PAF patients who underwent ablation procedure using the THERMOCOOL STSF Catheter as their first rhythm control therapy. The study will include consecutive, eligible patients from the REAL AF registry, starting from October 2021, who meet the sub-study eligibility criteria until 344 eligible subjects are identified.
  Eligible patients from all participating centers in the REAL AF registry will be included, except for sites with standard-of-care rhythm monitoring less than 48 hours, and those that do not perform 6-12 months follow-up as standard-of-care.
Sampling Method: Non-Probability Sample
Enrollment: 344 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Primary effectiveness | 12-months
  Freedom from atrial arrhythmia recurrence
Primary effectiveness | Post 3-month blanking period
  Any repeat ablation procedure, use of class I/III AAD, or cardioversion post-blanking for treatment of atrial arrhythmia will be deemed failure of primary effectiveness endpoint.
Primary safety | 7 days
  A composite of procedure or device related adverse events post index ablation.
Primary safety | 90 days
  Atrio-esophageal fistula, severe pulmonary vein stenosis and device or procedure related death post index ablation
Primary safety | 30 days
  Cardiac tamponade/pericardial effusion post index ablation

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Arrhythmia Institute at Grandview, Birmingham, Alabama
  - Community Memorial Hospital, Ventura, California
  - Ascension St. Vincent's, Jacksonville, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Northshore University Health System, Evanston, Illinois
  - Ascension St. Vincent's Hospital, Indianapolis, Indiana
  - Michigan Heart, Ypsilanti, Michigan
  - Mount Carmel Columbus Cardiology Consultants, Columbus, Ohio
  - University of Pennsylvania, Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Upstate Cardiology, Greenville, South Carolina
  - Centra Health, Inc. (dba Stroobants Cardiovascular Center), Lynchburg, Virginia